CLINICAL TRIAL: NCT03012386
Title: Role of CD36 in Nutrient Delivery and Its Dysfunction in African Americans
Brief Title: CD36 in Nutrient Delivery and Its Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 160955
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Insulin Resistance; Endothelial Dysfunction
Keywords: CD36; Endothelial dysfunction; African Americans
MeSH Terms: conditions — Insulin Resistance | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sildenafil citrate (Experimental): Sildenafil citrate 20 mg three times a day
  Interventions: Drug: Sildenafil Citrate in G allele carrier; Drug: Sildenafil Citrate in non G allele carrier

INTERVENTIONS:
Drug: Sildenafil Citrate in G allele carrier — chronic use of phosphodiesterase 5 inhibitor in G allele carrier
  Other Names: viagra, revatio,
Drug: Sildenafil Citrate in non G allele carrier — chronic use of phosphodiesterase 5 inhibitor in Non G allele carrier
  Other Names: viagra, revatio

SUMMARY:
This proposal will test the hypothesis that chronic treatment with sildenafil with and without the use of nitric oxide substrate, L-arginine, protects against fatty acid induced impairment of endothelial function, improves insulin-stimulated microvascular recruitment, insulin sensitivity and glucose uptake in CD36 rs3211938 G-allele carriers.

DETAILED DESCRIPTION:
Subjects carrying the G-allele of CD36 coding SNP rs3211938 that results in 50% reduction of CD36 levels in ~25% of African Americans have endothelial dysfunction. Endothelial dysfunction results in impairment of insulin's vascular actions and eventually reduced insulin sensitivity. Insulin induces microvascular recruitment via stimulation of nitric oxide(NO)-cGMP pathway, which facilitates nutrient flux, e.g., glucose to skeletal muscle. Elevated fatty acids impair insulin-stimulated microvascular recruitment and reduce insulin sensitivity. Chronic treatment with sildenafil increases vascularity and muscle glucose uptake in high fat fed mice. In humans, Drs. Shibao (PI) recently reported that a 3-month treatment with sildenafil improves insulin sensitivity in patients with impaired glucose tolerance. More relevant to this project, endothelial dysfunction improved after 4-week treatment with sildenafil in G-allele carriers. This proposal will test the hypothesis that chronic treatment with sildenafil with and without the use of NO substrate, L-arginine, protects against fatty acids induced impairment of endothelial function, improves insulin-stimulated microvascular.

The protocol design was changed to single arm design.

ELIGIBILITY:
Inclusion criteria

* African American men and women.
* Age 18-50 years
* BMI 25-40 kg/m2

Exclusion criteria:

* Diabetes type 1 or type 2, as defined by a FPG > 126 mg/dL a two-hour plasma glucose > 200 mg/dL, or the use of anti-diabetic medication
* Pulmonary hypertension
* Use of a PDE5 inhibitor for erectile dysfunction
* Pregnancy or breast-feeding. Women of child-bearing potential will be required to have undergone tubal ligation or to be using an oral contraceptive or barrier methods of birth control.
* Cardiovascular disease such as myocardial infarction, presence of angina pectoris, significant arrhythmia, congestive heart failure (left ventricular hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
* History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack
* History or presence of immunological or hematological disorders
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
* History of alcohol or drug abuse
* Mental conditions rendering a subject unable to understand the nature, scope and possible consequences of the study
* Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, unlikelihood of completing the study, and investigator discretion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shibao CA, Peche VS, Pietka TA, Samovski D, Williams IM, Abumrad NN, Gamazon ER, Goldberg IJ, Wasserman DH, Abumrad NA. Microvascular insulin resistance with enhanced muscle glucose disposal in CD36 deficiency. Diabetologia. 2025 Mar;68(3):662-675. doi: 10.1007/s00125-024-06292-4. Epub 2024 Nov 6. PMID 39503770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 subjects were screened, 9 were excluded for not meeting the inclusion criteria
Pre-assignment Details: 21 subjects completed the study
Groups:
- Sildenafil Citrate in G Allele Carriers; Sildenafil Citrate in Non Carriers of G Allele: Sildenafil citrate 20 mg three times a day
  Sildenafil Citrate: phosphodiesterase 5 inhibitor
Period: Overall Study
Arm/Group | Sildenafil Citrate in G Allele Carriers | Sildenafil Citrate in Non Carriers of G Allele
Started | 8 | 18
Completed | 8 | 13
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil Citrate in G Allele Carriers | Sildenafil Citrate in Non Carriers of G Allele | Total
Number analyzed (Participants) | 8 | 18 | 26
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 42 (7.4) | 33.66 (7.4) | 37.83 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 5 | 4 | 9
  Gender: Male | 3 | 14 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 18 | 26
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 169 (9.3) | 166.22 (8.72) | 167.61 (9.3)
Weight [Mean (Standard Deviation); unit: Kg] | 79 (8.34) | 92.95 (14.8) | 85.9 (14.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (2.8) | 33.53 (3.9) | 30.615 (3.9)
Glucose [Mean (Standard Deviation); unit: mg/dl] | 81 (10.0) | 83.5 (17.7) | 82.25 (17.7)
Total cholesterol [Mean (Standard Deviation); unit: mg/dl] | 180 (37.1) | 171.66 (29.48) | 175.83 (33.2)
HDL [Mean (Standard Deviation); unit: mg/dl] | 51 (13.8) | 53.38 (13.3) | 52.1 (13.6)
LDL [Mean (Standard Deviation); unit: mg/dl] | 106 (36.2) | 100.88 (28.25) | 103.44 (32.2)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 116.37 (73.85) | 87.11 (47.42) | 101.74 (60.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Microvascular Blood Volume (MBV) During Insulin Infusion
Description: Insulin induces microvascular recruitment. Changes in MBV during Insulin infusion signifies insulin sensitivity.
  MBV is measured in the forearm brachioradialis muscle with contrast enhanced ultrasonography during minutes 120-150 of a hyperinsulinaemic euglycaemic (HIE) clamp (insulin infusion rate up to 80 mU/m2.min-1 ). In the last 30 minutes, L-arginine was infused (10 mg/kg/min for 30 minutes) and ultrasound measurements were repeated upon infusion completion (approximately minute 180).
Time Frame: Baseline to end of procedure (approximately 180 minutes)
Measure: Mean (Standard Deviation); unit: ml/kg
Groups:
- G Allele Carriers: The participants were divided into two groups based on the CD36 rs3211938 genotype.
  subjects carrying the G-allele of CD36 coding SNP rs3211938 that results in reduction of CD36 levels
- Non Carriers of G Allele: The participants were divided into two groups based on the CD36 rs3211938 genotype.
Arm/Group | G Allele Carriers | Non Carriers of G Allele
Number analyzed (Participants) | 8 | 13
ml/kg | 13.16 (3.369) | 11.3 (1.37)

2. Primary Outcome: Change in Microvascular Blood Volume (MBV) During Insulin Infusion After 4 Weeks of Sildenafil Treatment in Both Groups
Description: Chronic treatment with sildenafil increases vascularity and muscle glucose uptake. Changes in MBV during Insulin infusion signifies insulin sensitivity .
  Insulin sensitivity was tested after 4 weeks of treatment with Sildenafil in both groups. Subjects receive IV infusion of 20% Intralipid (45ml/h) and heparin (200 units/hr). MBV is measured in the forearm brachioradialis muscle with contrast enhanced ultrasonography during minutes 120-150 of a HIE clamp (insulin infusion rate up to 80 mU/m2.min-1 ) In the last 30 minutes, L-arginine was infused (10 mg/kg/min for 30 minutes) and ultrasound measurements were repeated upon infusion completion (approximately minute 180).
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: ml/kg
Groups:
- Sildenafil Citrate in G Allele Carriers: Chronic use of phosphodiesterase 5 inhibitor in G allele carrier
  Other names: Viagra, Revatio
  Sildenafil citrate 20 mg three times a day for 4 weeks
- Sildenafil Citrate in Non Carriers of G Allele: Chronic use of phosphodiesterase 5 inhibitor in Non carriers of G allele
  Other names: Viagra, Revatio
  Sildenafil citrate 20 mg three times a day for 4 weeks
Arm/Group | Sildenafil Citrate in G Allele Carriers | Sildenafil Citrate in Non Carriers of G Allele
Number analyzed (Participants) | 8 | 13
ml/kg | 12.93 (2.31) | 8.4 (0.63)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Sildenafil Citrate
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 7/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil Citrate (N=26)
Positive pregnancy test (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Volunteer was terminated from the study due to positive and urine pregnancy tests
Malaria (Infections and infestations) | 1 (1) — non drug related event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil Citrate (N=26)
Rash and itchiness all over the body (Skin and subcutaneous tissue disorders) | 2 — Rash and pruritis was drug related. Subject responded to Hydroxyzine. No shortness of breath , no swelling and no wheezing was noted during the entire episode
Cough congestion (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1 — Diarrhea frst 5 days of taking study medication
Upset stomach / stomach virus (Infections and infestations) | 1
Burst of enerygy/ Irritability (Psychiatric disorders) | 1
Headaches (Nervous system disorders) | 3
Low back pain/ Leg heaviness (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT03012386/Prot_SAP_000.pdf